CLINICAL TRIAL: NCT05537558
Title: Toward PrecisiOn Medicine for the Prediction of Treatment Response in Major Depressive Disorder Through Stratification of Combined Clinical And-omics Signatures (PROMPT)
Brief Title: Precision Medicine for the Prediction of Treatment (PROMPT) Response (PROMPT)
Acronym: PROMPT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: University of Cagliari (Other); Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Bernhard Baune, Professor, University Hospital Muenster
Other Study IDs: University_of_Muenster_PROMPT
Record Dates: First submitted 2022-08-30; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Antidepressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antidepressant — Antidepressant (AD) monotherapy or complex psychopharmacology such as two ADs or AD plus augmentation (second generation antipsychotics, mood stabilizers, lithium, FT3/FT4). Combination with diverse types of ongoing psychotherapy will be accepted, if commenced prior to baseline

SUMMARY:
Major depressive disorder (MDD) is the most common psychiatric disease worldwide with a huge socio-economic impact. Pharmacotherapy represents the first-line treatment choice; however, only about one third of patients respond to the first trial and about 30% are classified as treatment-resistant depression (TRD). TRD is associated with specific clinical features and genetic/gene expression signatures. To date, single sets of markers have shown limited power in response prediction. The aim of this project is the development of a precision medicine algorithm that would help early detection of non-responder patients, who might be more prone to later develop TRD.

In this phase of the project a naturalistic cohort of 300 MDD patients will be recruited. The data collected will be used to assess, in real-world conditions, the capability of an innovative algorithm (integrating clinical, omics and gender data of other 300 patients con MDD) to predict the treatment outcomes. This project represents a proof-of-concept study. The obtained results will provide information about the feasibility and usefulness of the proposed approach, with the perspective of designing future clinical trials in which algorithms could be tested as a predictive tool to drive decision making by clinicians, enabling a better prevention and management of MDD resistance.

ELIGIBILITY:
Inclusion Criteria:

* A current diagnosis of moderate to severe MDD according to the DSM-IV was confirmed using the SCID-I diagnostic scale

Exclusion Criteria:

* Mental retardation or cognitive disorder
* A lifetime history of schizophrenic, schizoaffective, or bipolar disorder Substance abuse in the last 3 months
* Personality disorders, substance abuse, alcohol abuse, obsessive compulsive disorder, post-traumatic stress disorder, as primary diagnosis
* Comorbidity with eating disorders
* Substance or alcohol dependence

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: MDD in-patients or out-patients referred to psychiatric services are voluntarily enrolling in the study
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-09-09 (Estimated); Study Completion 2024-01-09 (Estimated)

PRIMARY OUTCOMES:
Clinical response | Baseline to 8 weeks
  Symptom improvement as measured by the percent change in the Montgomery-Asberg Depression Rating Scale (MADRS) score

SECONDARY OUTCOMES:
Clinical response and remission | Baseline to 2 weeks, to 4 weeks, to 8 weeks and 12 weeks
  Symptom improvement as well as response and remission rates as according to the MADRS

OTHER OUTCOMES:
Clinical response and remission self-reported | Baseline to 2 weeks, to 4 weeks, to 8 weeks and 12 weeks
  Changes in scores of depressive symptoms as measured by the Beck Depression Inventory II (BDI-II). Score on the BDI-II can range from 0 to 63 with higher scores indicating greater severity of depression.
Clinical response and remission self-reported | Baseline to 2 weeks, to 4 weeks, to 8 weeks and 12 weeks
  Changes in scores of anxiety symptoms as measured by the Beck Anxiety Inventory (BAI). Score on the BAI can range from 0 to 63 with higher scores indicating higher level of anxiety.
Psychosocial functioning | Baseline to 4 weeks, to 8 weeks and 12 weeks
  Changes in scores of psychosocial functioning as measured by the Functioning Assessment Short Test 24 items (FAST). All of items are rated using a 4-point scale. The global score is obtained when the scores of each item are added up. The higher the score, the more serious the difficulties are.
Side effects | Baseline to 4 weeks, to 8 weeks and 12 weeks
  Changes in side effects assessed by the UKU Side Effect Rating Scale (UKU-SERS). All of items are rated using a 3-point scale. Score can range from 0 to 63 with higher scores indicating more side effects.
Suicidal risk | Baseline to 2 weeks, to 4 weeks, to 8 weeks and 12 weeks
  Changes in scores of suicidal risk as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS). Scores on the C-SSRS can range from 0 to 25 with higher scores indicating higher intensity of suicidal risk. Anyway any score greater than 0 is important and may indicate the need for mental health intervention. The suicidal behavior lethality rating is taken directly from the C-SSRS.
Perceived stress | Baseline to 4 weeks, to 8 weeks and 12 weeks
  Changes in scores of perceived stress as measured by the Perceived Stress Scale-10 (PSS-10). Individual scores on the PSS-10 can range from 0 to 40 with higher scores indicating higher perceived stress.
General Health and Quality of Life | Baseline to 4 weeks, to 8 weeks and 12 weeks
  Changes in scores of quality of life as measured by the Quality of Life Questionnaire (SF-36). Consisting of 8 domains. The scores for each domain range from 0 to 100, with higher scores indicating more favorable health status.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard T. Baune, Professor, Principal Investigator — University Hospital Muenster
Locations (1):
- Bernhard Baune, Münster, Germany

IPD SHARING:
Plan to Share IPD: Undecided